CLINICAL TRIAL: NCT01151046
Title: A Randomized Double-Blind Phase 2 Trial of Exemestane +/- MM-121 in Postmenopausal Women With Locally Advanced or Metastatic Estrogen Receptor Positive (ER+) and/or Progesterone Receptor Positive (PR+) Her2 Negative Breast Cancer
Brief Title: Trial of Exemestane +/- MM-121 in Postmenopausal Women With Locally Advanced or Metastatic Estrogen Receptor Positive and/or Progesterone Receptor Positive Her2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MM-121-02-02-03 (ARD11588)
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Her2 Negative Breast Cancer Patients
Keywords: Breast Cancer; Her2 negative; Estrogen Receptor Positive; Progesterone Receptor Positive; MM-121; Exemestane; Postmenopausal Women
MeSH Terms: conditions — Breast Neoplasms | interventions — seribantumab; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MM-121 (SAR256212) + exemestane (Experimental)
  Interventions: Drug: MM-121; Drug: Exemestane
- Placebo + exemestane (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Exemestane

INTERVENTIONS:
Drug: MM-121 — MM-121 (40mg/kg loading dose week 1, then 20 mg/kg weekly) administered over 60 minutes as an intravenous infusion once per week
  Other Names: SAR256212
  Arms: MM-121 (SAR256212) + exemestane
Drug: Placebo — Placebo (histidine solution) administered over 60 minutes as an intravenous infusion once per week and exemestane (25 mg) administered orally once per day
  Arms: Placebo + exemestane
Drug: Exemestane — Exemestane (25 mg) administered orally once per day
  Other Names: Aromasin

SUMMARY:
To determine whether the combination MM-121 + Exemestane in ER+ and/or PR+ breast cancer patients is more effective than Exemestane alone

DETAILED DESCRIPTION:
The study is a double-blind, randomized Phase 2 trial of Exemestane +/- MM-121. The trial is designed to demonstrate whether MM-121 + Exemestane is more effective than Exemestane alone in ER+ and/or PR+ and Her2 negative breast cancer patients that have failed first-line anti-estrogen therapy in the locally advanced or metastatic setting and patients that have progressed during (or within 6 months of completing) adjuvant treatment with a non-steroidal aromatase inhibitor (AI)and/or tamoxifen. Patients will be treated until radiologic or clinical progression of their disease is documented. Local radiologist and/or PI assessment is accepted.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic breast cancer
* Histologically or cytologically confirmed ER+ and/or PgR+ and Her2 negative breast cancer
* ≥ 18 years of age

Exclusion Criteria:

* Received prior treatment with exemestane
* Extensive visceral disease (rapidly progressive, life-threatening metastases, including symptomatic lymphangitic metastases)
* Symptomatic CNS disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Moyo, MD, Study Director — Merrimack Pharmaceuticals, Inc.
Locations (32):
- United States (17):
  - Achieve Clinical Research, Birmingham, Alabama
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Pacific Cancer Medical Center, Anaheim, California
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Wilshire Oncology Medical Group, Inc., Corona, California
  - Southwest Cancer Center, Escondido, California
  - Hematology Oncology Associates, INC., Oakland, California
  - San Jose Medical Center, San Jose, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Pasco-Pinellas Oncology, New Port Richey, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tennessee Cancer Specialists Oncology Clinical Trials Center for Biomedical Research, Knoxville, Tennessee
  - Tennessee Cancer Specialists, Oncology Clincial Trials Center for Biomedical Research, Knoxville, Tennessee
- Canada (4):
  - Hopital Maissoneuve-Rosemont, Montreal, Quebec
  - McGill University Jewish General Hospital, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal
  - CHA St. Sacrement, Québec
- Germany (2):
  - Onkogologisches zentrum Munich, Munich
  - Brustzentrum HS Kliniken Wiesbaden, Wiesbaden
- Russia (4):
  - Medico-Diagnostically Center of International Institution of biological systems n.a.S.M., Berezina
  - Railway Clinical Hospital, Saint Petersburg
  - Leningrad Regional Oncology Center, Saint Petersburg
  - City Clinical Oncology Center, Saint Petersburg
- Spain (5):
  - Vall d'Hebrón University Hospital, Barcelona
  - Hospital Clinic (Barcelona), Barcelona
  - Hospital Parc Tauli - Barcelona, Barcelona
  - Servicio de Oncología Médica / Hospital Universitario Gregorio Marañón, Madrid
  - Puerta de Hierro, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- MM-121 + Exemestane: MM-121 (40mg/kg loading dose week 1, then 20 mg/kg weekly) administered over 60 minutes as an intravenous infusion once per week, plus exemestane (25 mg) administered orally once per day
- Placebo + Exemestane: Placebo and Exemestane: Placebo (histidine solution) administered over 60 minutes as an intravenous infusion once per week plus exemestane (25 mg) administered orally once per day
Period: Overall Study
Arm/Group | MM-121 + Exemestane | Placebo + Exemestane
Started | 59 | 59
Completed | 56 | 59
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- MM-121 + Exemestane: MM-121 and Exemestane: MM-121 (40mg/kg loading dose week 1, then 20 mg/kg weekly) administered over 60 minutes as an intravenous infusion once per week plus exemestane (25 mg) administered orally once per day
- Total: Total of all reporting groups
Arm/Group | MM-121 + Exemestane | Placebo + Exemestane | Total
Number analyzed (Participants) | 56 | 59 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 41 | 74
  >=65 years | 23 | 18 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.43) | 60.5 (9.13) | 61.6 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 59 | 115
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 55 | 56 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 2 | 0 | 2
  White | 54 | 57 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Bone-Only Disease (Y/N) [Number; unit: participants]
  Bone-Only (Yes) | 12 | 17 | 29
  Bone-Only (No) | 44 | 42 | 86
Progression Setting (Adjuvant, Metastatic) [Number; unit: participants]
  Adjuvant | 22 | 22 | 44
  Metastatic | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: To determine whether MM-121 + exemestane was more effective than placebo + exemestane in prolonging progression-free survival. PFS was a time to event measure, and progression of disease is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), "as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions". Progression free survival was defined as the number of months from the date of randomization to the date of death or progression. If neither death nor progression was observed during the study, PFS data was censored at the last non-progressive disease valid tumor assessment unless the patient was discontinued due to symptomatic deterioration. If this occurred, the patient was counted as having progressive disease (PD).
Time Frame: Time from first dose to date of progression, the longest time frame of 79.1 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MM-121 + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 56 | 59
weeks | 15.9 [9.3 to 30.3] | 10.7 [8.1 to 16.1]

2. Post Hoc Outcome: To Explore the Utility of an EGFR Family Receptor-ligand (Heregulin, HRG) as a Predictor of Response to MM-121 and /or Exemestane in Formalin Fixed (FFPE) Tumor Samples
Description: Fresh tumor samples were obtained from patients prior to enrollment and formalin-fixed for analysis. Samples were analyzed using RT-PCR for the expression of the biomarker, heregulin. Progression-free survival was assessed using RECIST v 1.1 to determine whether patients whose tumors express HRG have a lower PFS than those whose tumors do not express HRG, and to assess whether the addition of MM-121 to exemestane can increase PFS in HRG-high patients.
Time Frame: Time from first dose to date of progression, the longest time frame of 79.1 weeks
Population: Patients with available tissue for RT-PCR analysis
Measure: Median (95% Confidence Interval); unit: months PFS
Groups:
- HRG High: MM-121 + Exemestane; HRG Low: MM-121 + Exemestane: MM-121 (40mg/kg loading dose week 1, then 20 mg/kg weekly) administered over 60 minutes as an intravenous infusion once per week, plus exemestane (25 mg) administered orally once per day
- HRG High: Placebo + Exemestane; HRG Low: Placebo + Exemestane: Placebo and Exemestane: Placebo (histidine solution) administered over 60 minutes as an intravenous infusion once per week plus exemestane (25 mg) administered orally once per day
Arm/Group | HRG High: MM-121 + Exemestane | HRG High: Placebo + Exemestane | HRG Low: Placebo + Exemestane | HRG Low: MM-121 + Exemestane
Number analyzed (Participants) | 16 | 18 | 19 | 23
months PFS | 3.8 [1.9 to NA] — Confidence interval upper limit not reached | 1.9 [1.8 to 3.6] | 5.4 [1.9 to NA] — Confidence interval upper limit not reached | 3.5 [1.7 to NA] — Confidence interval upper limit not reached
Statistical Analysis 1: Comparison: HRG High: MM-121 + Exemestane vs HRG High: Placebo + Exemestane; Test type: Superiority or Other; p = 0.003, Log Rank; Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.11 to 0.63]
Statistical Analysis 2: Comparison: HRG Low: Placebo + Exemestane vs HRG Low: MM-121 + Exemestane; Test type: Superiority or Other; p = 0.349, Log Rank; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.69 to 2.88]

3. Secondary Outcome: Overall Survival
Description: To determine whether MM-121 + exemestane is more effective than placebo + exemestane in prolonging overall survival. This was a time-to-event analysis of time from first dose to date of death.
Time Frame: Time from first dose to date of death, over approximately 2 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MM-121 + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 56 | 59
weeks | NA [NA to NA] — endpoint was not reached. | 96.3 [51.4 to 96.3]

ADVERSE EVENTS:
Time Frame: AEs were collected from a patient's first dose until 30 days after treatment termination. SAEs were collected from time of informed consent until 30 days after termination. If related, events could be reported at any time after termination.
Description: All related AEs ongoing at treatment discontinuation were followed until resolution. Investigators were to report any AEs/SAEs assumed to be related any time, even if occurring more than 30 days after last dose. Though different for each patient, on average, patients could be followed for related AEs/SAEs for up to 2 years after termination.
Arm/Group | MM-121 + Exemestane | Placebo + Exemestane
Serious Adverse Events (participants affected / at risk) | 7/56 | 11/59
Other Adverse Events (participants affected / at risk) | 48/56 | 50/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MM-121 + Exemestane (N=56) | Placebo + Exemestane (N=59)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Tacchycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Upper) (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 1 (1) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (General disorders) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Horner's Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MM-121 + Exemestane (N=56) | Placebo + Exemestane (N=59)
Diarrhea (Gastrointestinal disorders) | 28 | 14
Nausea (Gastrointestinal disorders) | 16 | 14
Fatigue (General disorders) | 13 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Decreased Appetite (Metabolism and nutrition disorders) | 9 | 5
Dysgeusia (Nervous system disorders) | 8 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 6
Aspartate Aminotransferase Increased (Investigations) | 7 | 3
Asthenia (General disorders) | 7 | 6
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 0
Headache (Nervous system disorders) | 7 | 12
Insomnia (Psychiatric disorders) | 7 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 6 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 9
Constipation (Gastrointestinal disorders) | 6 | 5
Dizziness (Nervous system disorders) | 6 | 6
Stomatatitis (Gastrointestinal disorders) | 6 | 1
Alanine Aminotransferase Increased (Investigations) | 5 | 2
Hypokalemia (Metabolism and nutrition disorders) | 5 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 5 | 9
Abdominal Pain (Gastrointestinal disorders) | 4 | 4
Anemia (Blood and lymphatic system disorders) | 4 | 7
Influenza-like illness (General disorders) | 4 | 3
Peripheral edema (General disorders) | 4 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 6
Pyrexia (General disorders) | 4 | 4
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 3
Urinary Tract Infection (Infections and infestations) | 4 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 3 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Cellulitis (Infections and infestations) | 3 | 1
Chest Pain (General disorders) | 3 | 0
Dry Eye (Eye disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 7
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hot Flush (General disorders) | 3 | 7
Influenza (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 3 | 3
Parasthesia (Nervous system disorders) | 3 | 3
Pollakuria (Renal and urinary disorders) | 3 | 2
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 3 | 0
Weight Decreased (Investigations) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no overall study publication has occurred by the Sponsor within 12 months of the completion of this Study, the Investigator shall have the right to publish or present independently the results of this Study subject to the review procedure set forth herein. The Investigator will provide the Sponsor with a copy of any such presentation or publication derived from the Study for review, and the Sponsor may delay publication for up to 90 days to preserve patent activities and proprietary rights.